CLINICAL TRIAL: NCT07164404
Title: Increasing Nicotine Replacement Therapy Prescribing and Lung Cancer Screening in Hospitalized Patients Using an Innovative Non-Interruptive Alert Within the Electronic Health Record Provider Note
Brief Title: Nicotine Replacement Therapy Prescribing and Lung Cancer Screening in Hospitalized Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: South Carolina Clinical & Translational Research Institute (SCTR) (Unknown)
Responsible Party: Principal Investigator, Ellen Esposito, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00146588
Record Dates: First submitted 2025-08-28; First posted 2025-09-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EHR alert (Experimental): Group will have access to the EHR embedded alert into the admission note template, where it automatically inserts smoking history, prompts NRT prescribing in the hospital, and offers referral to outpatient follow up.
  Interventions: Other: EHR alert
- Control (No Intervention): Routine care, no access to the EHR embedded alert

INTERVENTIONS:
Other: EHR alert — EHR embedded alert into the admission note template, where it automatically inserts smoking history, prompts NRT prescribing in the hospital, and offers referral to outpatient follow up.
  Arms: EHR alert

SUMMARY:
Investigators are evaluating an EHR-based, non-interruptive alert to increase NRT prescribing in the hospital and at discharge for hospitalized patients. Investigators will investigate two randomized groups of resident physicians to evaluate their prescribing behaviors when the tool is introduced.

DETAILED DESCRIPTION:
Efforts to decrease cancer-related morbidity and mortality include increasing smoking cessation, however smoking remains prevalent. Classically, alerts within the electronic health record (EHR) are implemented to address gaps in care, yet studies suggest typical EHR alerts are often overridden and ignored. In this study, the investigators aim to decrease the incidence and burden of disease by including hospitalists as part of the multidisciplinary care team by implementing and evaluating a novel non-interruptive EHR alert embedded within a provider note as a tool to increase prescription of nicotine replacement therapy to patients who smoke upon admission to and discharge from the hospital. Investigators will investigate two randomized groups of resident physicians to evaluate their prescribing behaviors when the tool is introduced.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Hospitalized patients admitted to a General Medicine Service at MUSC Charleston
* Identified as actively smoking tobacco via nursing admission screening
* Admitted by a resident physician participating in the study (as indicated by the H&P note)

Exclusion Criteria:

• None

Resident Physicians:

Inclusion Criteria:

• Internal medicine resident physicians rotating on the hospitalist service at MUSC Health Charleston

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Nicotine Replacement Therapy (NRT) prescribing rates during hospitalization | During hospitalization, assessed from admission to discharge (average of 3-7 days)
Nicotine Replacement Therapy (NRT) prescribing rates at discharge | During hospitalization, assessed from admission to discharge (average of 3-7 days)
Rate of referral to outpatient tobacco cessation clinic | During hospitalization, assessed from admission to discharge (average of 3-7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Esposito, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No